CLINICAL TRIAL: NCT01882738
Title: Effect of Maternal BMI on Accuracy of Measurement of Cervical Length During the 3rd Trimester of Pregnancy
Brief Title: Effect of Maternal BMI on Measurement of Cervical Length
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0039-13-HYMC
Record Dates: First submitted 2013-06-11; First posted 2013-06-20 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: PREGNANCY
Keywords: Cervical length; BMI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
All consecutive pregnant patients in 2nd or 3rd trimester will be asked to participate. Cervical length will be assessed in all patients, once abdominally and then vaginally (that would serve as golden standard). Correlation would be assessed between accuracy of measurement to BMI

DETAILED DESCRIPTION:
This study will include pregnant women in either 2nd or 3rd trimester of pregnancy. All consecutive pregnant patients in 2nd or 3rd trimester who will attend our unit for routine ultrasound exam will be asked to participate. Cervical length will be assessed in all patients, once abdominally and then vaginally (that would serve as golden standard). Correlation would be assessed between accuracy of measurement to BMI. Accuracy would be defind as the delta of cervical length between abdominal and vaginal routs.

BMI would be calculated prior to the ultrasound exam (by weighing and measuring all patients).

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women in 2nd or 3rd trimester who attend routine ultrasound exam

Exclusion Criteria:

* Known shore cervix
* PPROM

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All pregnant women in 2nd or 3rd trimester who attend routine ultrasound exam
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Accuracy of cervical length according to BMI | 1 year
  the golden standard for cervical length measurement is vaginal scan. Our outcome measure will be the accuracy of cervical length measurement - measured abdominally, according to BMI. I other words - was there a difference between measurement by vaginal probe and abdominal probe and whether this difference correlates with BMI

SECONDARY OUTCOMES:
Gestational age at delivery according to cervical length | 1 year
  Gestational age at delivery according to cervical length

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel